CLINICAL TRIAL: NCT00166387
Title: Hemophilia Inhibitor Genetics Study (HIGS)
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Sharyne M. Donfield, Ph.D., Professor Erik Berntorp, Malmö University Hospital, Skane University Hospital
Other Study IDs: HIGS
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Hemophilia A With Inhibitor
Keywords: Hemophilia; Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based
Biospecimen Retention: Samples With DNA — Plasma, cells, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Phase I, II, III: Phase I consists of a brother pair with hemophilia, one or both of whom has a history of inhibitors, and their parents; Phase II consists of a person with hemophilia and an inhibitor, and both his parents; Phase III consists of an unrelated group of people with hemophilia.
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — A single blood draw.
  Other Names: N/A to this study.

SUMMARY:
Several non-genetic and genetic factors that could influence the risk of inhibitor development in hemophilia A have been discussed but not fully explored. The aim of the HIGS is to identify these genetic factors.

DETAILED DESCRIPTION:
The objective of the HIGS is to determine host genetic factors, other than mutations within the factor VIII gene, that are associated with the development of inhibitors in severe hemophilia A and response to antigenic challenge by factor VIII. The study will involve three phases, enrolling family groups composed of brother pairs and their parents (Phase I) and siblings, a family group composed of a person with severe hemophilia and his parents (Phase II), and a group of unrelated people with severe hemophilia for the purpose of confirming associations identified in Phases I and II.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A is defined as a baseline factor VIII level <1%. A history of inhibitor is defined as ever having a Bethesda titer > 1 BU.

Phase I.

Subjects with hemophilia are eligible for Phase I of the study if all of the following apply:

* An informed consent form, approved by the appropriate IRB/IEC, has been administered, signed, and dated.
* The subject has severe hemophilia A.
* The subject has a history of inhibitor or the subject has no history of inhibitor but has at least 100 exposure days to factor VIII products.
* Sufficient documentation exists to identify the subject's maximum lifetime Bethesda titer.
* The subject has a history of inhibitor and has one or more full brothers with severe hemophilia A, with or without an inhibitor, who are eligible for and have agreed to be in the study, and two parents who have agreed to be in the study or the subject does not have a history of inhibitor but has one or more full brothers with severe hemophilia A and a history of inhibitor who are eligible for and have agreed to be in the study, and two parents who have agreed to be in the study.

Subjects without hemophilia are eligible for Phase I of the study if all of the following apply:

* An informed consent form, approved by the appropriate IRB/IEC, has been administered, signed, and dated.
* The subject is the parent (mother or father) of, or the full sibling of, a subject with hemophilia who is eligible for Phase I of the study.

Phase II.

Subjects with hemophilia are eligible for Phase II of the study if all of the following apply:

* An informed consent form, approved by the appropriate IRB/IEC, has been administered, signed, and dated.
* The subject has severe hemophilia A.
* The subject has a history of inhibitor and two parents who have agreed to be in the study.
* Sufficient documentation exists to identify the subject's maximum lifetime Bethesda titer.

Subjects without hemophilia are eligible for Phase II of the study if all of the following apply:

* An informed consent form, approved by the appropriate IRB/IEC, has been administered, signed, and dated.
* The subject is the parent (mother or father) of a subject with hemophilia who is eligible for Phase II of the study.

Exclusion Criteria:

Phase I.

Subjects (with or without hemophilia) are excluded from participation in Phase I if:

* The minimum family group, defined as a pair of full brothers with hemophilia, either concordant (both with) or discordant (one with, one without) for inhibitor, and both of their parents, is not enrolled.

Phase II.

Subjects are excluded from participation in Phase II if:

* The minimum family group, defined as a person with hemophilia and a history of inhibitor and his mother and father, is not enrolled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with hemophilia and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 1137 (Actual)
Dates: Start 2003-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
development of inhibitory antibodies to factor VIII | upon development of inhibitor or following at least 100 exposure days to factor VIII

CONTACTS AND LOCATIONS:
Overall Officials: Erik Berntorp, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Malmo University Hospital, Malmo, Sweden

REFERENCES:
- [Background] Berntorp E, Astermark J, Donfield SM, Nelson GW, Oldenburg J, Shapiro AD, Dimichele DM, Ewenstein BM, Gomperts ED, Winkler CA; Hemophilia Inhibitor Genetics Study. Haemophilia Inhibitor Genetics Study - evaluation of a model for studies of complex diseases using linkage and association methods. Haemophilia. 2005 Jul;11(4):427-9. doi: 10.1111/j.1365-2516.2005.01119.x. No abstract available. PMID 16011603
- [Background] Astermark J, Donfield SM, Gomperts ED, Schwarz J, Menius ED, Pavlova A, Oldenburg J, Kessing B, DiMichele DM, Shapiro AD, Winkler CA, Berntorp E; Hemophilia Inhibitor Genetics Study (HIGS) Combined Cohort. The polygenic nature of inhibitors in hemophilia A: results from the Hemophilia Inhibitor Genetics Study (HIGS) Combined Cohort. Blood. 2013 Feb 21;121(8):1446-54. doi: 10.1182/blood-2012-06-434803. Epub 2012 Dec 6. PMID 23223434
- [Background] Schwarz J, Astermark J, Menius ED, Carrington M, Donfield SM, Gomperts ED, Nelson GW, Oldenburg J, Pavlova A, Shapiro AD, Winkler CA, Berntorp E; Hemophilia Inhibitor Genetics Study Combined Cohort. F8 haplotype and inhibitor risk: results from the Hemophilia Inhibitor Genetics Study (HIGS) Combined Cohort. Haemophilia. 2013 Jan;19(1):113-8. doi: 10.1111/hae.12004. Epub 2012 Sep 7. PMID 22958194